CLINICAL TRIAL: NCT01992991
Title: Transcranial Direct Current Stimulation for Upper Limb Training of Individuals With Sequelae From Intracranial Hemorrhage
Brief Title: Transcranial Stimulation for Upper Limb Training of Individuals With Sequelae From Intracranial Hemorrhage
Acronym: tDCS-ICH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCS-RHN
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Cerebrovascular Disorders
Keywords: transcranial stimulation; Intracranial hemorrhage; Home training; Occupational Therapy; Jebsen Taylor Hand Function Test
MeSH Terms: conditions — Cerebrovascular Disorders; Intracranial Hemorrhages | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial direct current stimulation (Experimental): Anodal stimulation
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): 30 sek of Transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation of motor cortex

SUMMARY:
The purpose of this study is to investigate the effect of transcranial stimulation for upper limb training of patients with sequelae from an intracranial hemorrhage.

Patients receive five days of upper limb occupational therapy training in combination with real or sham stimulation. Patients complete the Jebsen Taylor Hand Function Test before, after and 7 days later. The intervention takes place at patients' home address.

DETAILED DESCRIPTION:
Aim: To investigate the effect of anodal transcranial direct current stimulation (tDCS) for upper limb training of individuals with sequelae from intracranial hemorrhage.

Design: Triple-blinded randomised controlled trial Study population: Patients with intracranial hemorrhage (ICH) of non-traumatic aetiology. Between 6 months and five years from injury.

Intervention:

Group 1 receive five days of upper limb occupational therapy in combination with anodal stimulation Group 2 receive five days of upper limb occupational therapy in combination with sham stimulation The intervention takes place at patients' home address. Assessment tool: Patients complete the Jebsen Taylor Hand Function Test at baseline, post-intervention and at 7 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial hemorrhage
* Injury between 6 months and 5 years

Exclusion Criteria:

* Traumatic brain injury
* Other neurological disorders
* Epilepsy
* Metal implants in the head

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change in Jebsen Taylor Hand Function Test | Change from baseline until 7 days follow-up
  Involves seven items regarding activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD, PhD, Study Director — Hammel Neurorehabilitation and Research Centre
Locations (1):
- Hammel Neurorehabilitation and Research Centre, Hammel, Jutland, Denmark